CLINICAL TRIAL: NCT02355158
Title: A Multicenter, Open-label, Single-arm Study to Evaluate the Long-term Use of Clonidine Hydrochloride Topical Gel, 0.1% in the Treatment of Pain Associated With Painful Diabetic Neuropathy
Brief Title: A Safety Study of Clonidine Hydrochloride Topical Gel, 0.1% in the Treatment of Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioDelivery Sciences International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLO-311
Record Dates: First submitted 2014-11-21; First posted 2015-02-04 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-08

CONDITIONS: Painful Diabetic Neuropathy; Diabetes
Keywords: pain; diabetic neuropathy; pain in feet
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active (Experimental): Clonidine hydrochloride topical gel, 0.1%
  Interventions: Drug: clonidine hydrochloride topical gel, 0.1%

INTERVENTIONS:
Drug: clonidine hydrochloride topical gel, 0.1%

SUMMARY:
Study CLO-311 is a multicenter, open-label, single-arm study to assess the long-term use of Clonidine Gel in the treatment of pain associated with PDN. Subjects who have completed their 12-week participation in Study CLO-290 or Study CLO-310 are eligible to rollover into this study and receive active study drug in an open-label manner.

DETAILED DESCRIPTION:
Study CLO-311 is a multicenter, open-label, single-arm study to assess the long-term use of Clonidine Gel in the treatment of pain associated with PDN. Subjects who have completed their 12-week participation in Study CLO-290 or Study CLO-310 are eligible to rollover into this study and receive active study drug in an open-label manner. All eligible subjects will receive Clonidine Gel regardless of the blinded treatment they have received in the previous double-blind study (Clonidine Gel or Placebo Gel). Study drug will be applied topically TID to both feet for 12 months during an Open-Label Treatment Phase. Approximately 400 adult subjects with PDN are estimated to enroll in this study.

ELIGIBILITY:
Inclusion Criteria:

* The subject has provided written informed consent.
* The subject has Type 1 or Type 2 diabetes mellitus with glycemic control that has been optimized on diet therapy, oral anti-hyperglycemic agents and/or insulin.
* The subject must be a male or non-pregnant, non-lactating female. Females must be practicing an acceptable method of birth control, or be surgically sterile or postmenopausal (amenorrhea for ≥12 months). Non-pregnancy will be confirmed (as applicable) by a pregnancy test conducted at the Entry Visit. Double-barrier methods, hormonal contraceptives, and abstinence are acceptable birth control methods for this study.
* The subject has completed their 12-week participation according to the protocol in the previously conducted double-blind study, CLO-290.
* The subject is medically stable at the end-of-study visit (Day 85) of Study CLO-290, and in the opinion of the Investigator, is in otherwise good general health based on physical examination, ECG, and laboratory evaluation.
* Subject has the capabilities of applying topical gel to both feet TID. A caregiver, trained by the study staff to apply study medication, would be a suitable alternative to self-application of the treatment.

Exclusion Criteria:

* The subject is using an implanted medical device (e.g., spinal cord stimulator, intrathecal pump, or peripheral nerve stimulator) for the treatment of pain.
* The subject is clinically hypotensive with a resting diastolic blood pressure <60 mmHg or a systolic blood pressure <90 mmHg.
* The subject has recent history (within the past 3 months) or current symptoms of orthostatic hypotension with a sudden fall in blood pressure on standing accompanied by dizziness and lightheadedness.
* The subject has any significant or unstable medical or psychiatric condition that, in the opinion of the Investigator, would interfere with his/her ability to participate in the study.
* The subject has a history of substance abuse disorder as defined by DSM-IV-TR within the past 6 months, has current evidence for substance abuse disorder, or is receiving medicinal treatment for drug abuse.
* The subject has symptomatic or severe coronary insufficiency, clinically significant cardiac conduction disturbances, myocardial infarction (within last 6 months), cerebrovascular disease, or chronic obstructive pulmonary disease (COPD) requiring oxygen therapy.
* The subject is likely to be noncompliant or unreliable in providing ratings as judged by the Investigator.
* The subject has evidence of clinically significant peripheral vascular disease as evidenced by a history of intermittent claudication or evidence of vascular ulcers, including venous stasis ulcers.
* The subject is currently taking or has taken clonidine in any form other than Clonidine Gel study drug (i.e., oral, transdermal patch) over the past 4 months.
* The subject has developed hypersensitivity or intolerance to clonidine.
* The subject is currently receiving any non-oral treatment that could affect neuropathic pain.
* Subject has a history of malignancy within the past 5 years with the exception of successfully treated non-metastatic basal cell or squamous cell carcinomas of the skin and/or localized carcinoma in situ of the cervix.
* The subject has clinical evidence of pedal edema or venous stasis disease associated with significant skin changes on physical examination.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Shaibani, MD, Principal Investigator — Nerve & Muscle Center of Texas
Locations (19):
- United States (19):
  - Phoenix, Arizona
  - Santa Monica, California
  - Walnut Creek, California
  - Waterbury, Connecticut
  - Bradenton, Florida
  - Brandon, Florida
  - Jupiter, Florida
  - Miami, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Columbus, Georgia
  - Kansas City, Kansas
  - Hazelwood, Missouri
  - Winston-Salem, North Carolina
  - Warwick, Rhode Island
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Renton, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active
Started | 197
Completed | 47
Not Completed | 150

BASELINE CHARACTERISTICS:
Arm/Group | Active
Number analyzed (Participants) | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40
  Not Hispanic or Latino | 157
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 47
  White | 146
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 197

OUTCOME MEASURES:

1. Primary Outcome: Summary of Neuropathic Pain Symptom Inventory (NPSI)
Description: The NPSI is a validated, self-administered questionnaire designed to evaluate the different symptoms of neuropathic pain. Each item is quantified on an 11-point (0-10) numeric scale. The NPSI includes 10 descriptors (plus 2 temporal items) that allow discrimination and quantification of 5 distinct clinically relevant dimensions of neuropathic pain syndromes. The Neuropathic Pain Symptom Inventory (NPSI) is a self-questionnaire designed to evaluate the different symptoms of neuropathic pain, which contains a list of descriptors reflecting spontaneous ongoing or paroxysmal pain, evoked pain (i.e., mechanical and thermal allodynia/hyperalgesia) and dysesthesia/paresthesia. Each of these items is quantified on an 11-point (0-10) numerical scale. NPSI total score was calculated and summarized descriptively at month 12 or the subjects last visit. The total score was calculated and summarized.
Time Frame: Month 12 or last visit
Population: While 197 subjects received study drug, 172 completed the NPSI at the week 12 visit or at their last visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active
Number analyzed (Participants) | 172
units on a scale | 34.44 (25.13)

ADVERSE EVENTS:
Time Frame: 1 year 7 days
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE (also referred to as an adverse experience) may have been any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, without any judgment about causality.
Arm/Group | Active
All-Cause Mortality (participants affected / at risk) | 1/197
Serious Adverse Events (participants affected / at risk) | 23/197
Other Adverse Events (participants affected / at risk) | 79/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=197)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Myodcaridal infarction (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Ischaemic limb pain (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=197)
Upper respiratory tract infection (Infections and infestations) | 11 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (11)
Headache (Nervous system disorders) | 27 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days